CLINICAL TRIAL: NCT07026097
Title: Effects of Online Versus Physically Supervised Pilates Exercise Program With Common Standard Physical Therapy Treatment on Pain, Mobility and Function in Patients With Non-specific Low Back Pain
Brief Title: Online Versus Physically Supervised Pilates Exercise Program in Non-specific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Summya - REC/RCR&AHS 24/0138
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Pilates Training; Pilates Based Exercises; Range of Motion; Disability
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Pilates Exercise - Online
- Group B (Active Comparator)
  Interventions: Other: Pilates Exercise - Supervised

INTERVENTIONS:
Other: Pilates Exercise - Online — Will receive Pilates exercise protocol online under supervision as patient will instructed to join online meeting and do their exercise 02 times a week along with standard physical therapy protocol for 4 weeks. The Pilates exercise protocol will be of 30 minutes. Repetitions: Exercises started with 6 to 10 reps. and hold time for 30 sec for each exercise. Rest period of 2 mins will be given
  Arms: Group A
Other: Pilates Exercise - Supervised — Will receive Pilates exercise protocol clinically supervised as patient will instructed to do their exercise 0 times a week along with standard physical therapy protocol for 4 weeks. The Pilates and common standard physical therapy protocol will be the same which is mention in detail in group A description
  Arms: Group B

SUMMARY:
The study will be Randomized Controlled Trial and will be conducted in Riphah Rehabilitation Research Center. The study duration will be 9 months. Non- probability convenient sampling technique will be used to collect the data. Patients with chronic non-specific low back pain will be included in this study after meeting the inclusion criteria. The sample size of this study is 40 participants 20 in each group. Both groups will be an experimental group and will receive Pilates exercise protocol and common standard physical therapy treatment, 02 times a week for 04 weeks. Group A will receive supervised online Pilates exercise plan with common standard physical therapy and Group B will receive clinical supervised Pilates with common standard physical therapy treatment. The common standard physical therapy plan will be a hot pack for lumbar region for 10 mins, hamstring stretch, participants should maintain this stretch for 30 secs with 10 repetitions and strengthening of abdominal muscles in crook lying position with 10 repetitions with hold of 30 sec. The Pilates exercise protocol will include rollup, one leg circle exercise, crook leg lying, prone single leg kick, side-lying clamshell, supine stretch exercise, bug roll, prone attitude rotation, side kick and saw exercise. The Pilates protocol will be of 30 mins with 06-10 repetitions for each exercise withhold time for 30 sec. The outcome measure will be Numeric Pain Rating Scale (NPRS) for pain, Oswestry Low Back Disability Questionnaire (ODI) for disability and inclinometer for range of motion.

DETAILED DESCRIPTION:
Low back pain (LBP) is characterised by pain, muscle tension or stiffness located below the 12th rib and above the gluteal folds . In many patients, the specific nociceptive source of LBP cannot be identified and those affected are often classified as having nonspecific low back pain. Nonspecific LBP represents 90% to 95% of cases . Chronic non-specific LBP (CNLBP) is distinguished by persistent pain for more than 12 weeks, without a clear cause. This condition is considered one of the most common causes of disability. It is estimated that 80% of adults have at least one episode of LBP during their lifetime and aproximately 85% of cases falling under the umbrella of non-specific LBP, often labelled as idiopathic low back dysfunction due to the absence of identifiable anatomical abnormalities .

Low back pain (LBP) is a great public health issue and the second most common cause of seeking advice from a physician. It is the leading source of human suffering and disability worldwide . Approximately 15% to 20% of adults suffer from back pain each year. The issue is common in both developing and developed countries of the world . As compared to developed countries low back pain is more prevalent in developing countries. It is considered the second most common disease in adults under the age of 45 years .

The prevalence of low back pain among older population is 40.6% in Pakistan. In Pakistan, the prevalence is notably high, ranging from 29.20% to 70%. Individuals experiencing low back dysfunction grapple with various musculoskeletal symptoms, including pain, restricted range of motion (ROM) and a decline in functional indices. Now a days low back pain is also very common is younger population a study shows that 25.1% males and 36.8% females of age ranging 18-25 also experience low back pain in Pakistan. 84% population of USA have low back pain. it is estimated that 70-85% of the working population has suffered from a LBP episode, with many reports of long periods of absence from their jobs, restricting their physical activity and affecting their output and the quality of life.

With the rise of digital platforms and global pandemic, there has been a significant shift towards online fitness program. Investigating the effectiveness of online Pilates can provide information whether these programs will work better compared to traditional, in person programs. Online Pilates offers greater accessibility for individuals who, may not have an easy access to clinics due to geographic, financial or time constraints. This research will help determine if online Pilates can deliver similar benefits to in-person therapy, making treatment more accessible to patients. This study will help practitioners in making informed choices whether online Pilates or clinical Pilates which is better for the patients. Another impact is that by giving treatment online cost of the treatment will also reduce which is beneficial for the patients. So, the purpose of this study is to compare the effects of online versus physically supervised Pilates exercise program with common standard Physical Therapy Treatment on pain, mobility and function in patients with non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LBP
* Minimum chronicity of LBP 03
* Both Gender
* Age ranges from 18-40
* Numeric pain rating scale (NPRS) score 3 to 8 for pain intensity
* Patient who can maintain their standing posture independently for ≥30 minutes, have enough physical autonomy to participate in the physical activities required by the study
* Oswestry Disability Index score 20-34

Exclusion Criteria:

* History of trauma or fracture of the supine
* Chronic systemic soft tissue or bony disease
* Post Operative
* Pregnancy
* Diagnosis of osteoarthritis and herniated disc
* Any medical red flags
* Neurological and visual impairments
* Presence of root symptoms (e-g sciatica and cauda equina syndrome)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Baseline, 4th week
Oswetry Disability Index | Baseline, 4th week
Lumbar Range of Motion | Baseline, 4th week

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddiqui AS, Javed S, Abbasi S, Baig T, Afshan G. Association Between Low Back Pain and Body Mass Index in Pakistani Population: Analysis of the Software Bank Data. Cureus. 2022 Mar 30;14(3):e23645. doi: 10.7759/cureus.23645. eCollection 2022 Mar. PMID 35510015
- [Background] Nieminen LK, Pyysalo LM, Kankaanpaa MJ. Prognostic factors for pain chronicity in low back pain: a systematic review. Pain Rep. 2021 Apr 1;6(1):e919. doi: 10.1097/PR9.0000000000000919. eCollection 2021. PMID 33981936